CLINICAL TRIAL: NCT02288104
Title: Needle-based Confocal Laser Endomicroscopy in CT-guided Procedures in Interventional Radiology With Applications in Liver and Kidneys: a Feasibility Study
Brief Title: Needle-based Confocal Laser Endomicroscopy in CT-guided Percutaneous Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mauna Kea Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKT-IR-NHC-2014
Record Dates: First submitted 2014-10-27; First posted 2014-11-11 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Liver Percutaneous Biopsy or Ablation; Kidney Percutaneous Biopsy or Ablation
Keywords: Interventional Radiology; Liver; Kidney; Confocal endomicroscopy; Optical Biopsy; Scanner; Fluoroscopy; CT; Computed Tomography; Radiofrequency Ablation; Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- needle based confocal endomicroscopy (Other): The patient, scheduled for a standard liver or kidney percutaneous biopsy or ablation will undergo a needle-based confocal laser endomicroscopy procedure during the procedure. The objectives of this study are to demonstrate the technical feasibility and safety of doing endomicroscopic imaging during interventional radiology procedure and determine whether it is technically feasible to obtain images from Cellvizio during an interventional radiology procedure.
  Interventions: Device: needle based confocal endomicroscopy

INTERVENTIONS:
Device: needle based confocal endomicroscopy — real time imaging of living tissue at microscopic scale, through a needle.

SUMMARY:
This study is a prospective study in order to demonstrate the technical feasibility and safety of doing endomicroscopic imaging during interventional radiology procedure in two main indications: Kidneys and liver.

This innovative study will involve the use of probe-based confocal laser endomicroscopy. The proposed study is a feasibility study.

DETAILED DESCRIPTION:
Interventional radiology is a medical sub-specialty of radiology which utilizes minimally-invasive image-guided procedures to diagnose and treat diseases in nearly every organ. The concept behind interventional radiology is to diagnose and treat patients using less invasive techniques currently available in order to minimize risk to the patient and improve health outcomes.

For many years, surgery was the only treatment available for many conditions. Today, interventional radiology treatments are frst-line care for a wide variety of conditions. Patients should be offered the least invasive option frst. It is important to get a second opinion and know all of your treatment options before consenting to any procedure or surgery. Interventional radiologists are specialists in minimally invasive treatments, have a unique breadth of training and provide consults to every type of specialist.

Surgical removal of liver tumors offers the best chance for a cure. Unfortunately, liver tumors are often inoperable because the tumor may be too large, or has grown into major blood vessels or other vital structures. Sometimes, many small tumors are spread throughout the liver, making surgery too risky or impractical. Surgical removal is not possible for more than two-thirds of primary liver cancer patients and 90 percent of patients with secondary liver cancer.

The objectives of this study are to demonstrate the technical feasibility and safety of doing endomicroscopic imaging during interventional radiology procedure in two main indications: liver and kidneys.

The Primary objective is:

To study and demonstrate the technical feasibility and safety of doing endomicroscopic imaging during interventional radiology procedure in two main indications: liver and kidney.

The Secondary objectives are:

1. Assess the safety of the use of Endomicroscopic imaging during interventional radiology procedure in two main indications: liver and kidney.
2. Assess the quality of biopsies performed with the help of Cellvizio.
3. Build a database of images as an atlas and define image interpretation criteria in collaboration with pathologists.

Evaluate whether and how Cellvizio can improve guidance for biopsies or ablations: for instance, in the critical structures such as nerves or vessels in the vicinity of the cryoablation area, is it possible to visualize ice crystals and therefore decide to stop the cryoablation at the right time/location?

For both applications, technical feedback from the physicians is expected on how they think the combined use of the devices could change the care path. E.g. a certain step in the workflow might become obsolete or the workflow could lead to fewer patient visits.

For the safety of this protocol, the use of endomicroscopy will not change in any way the patient management and standard procedure, including the diagnosis nor treatment decisions. All the adverse events / serious adverse events will be noted during the procedure and one week after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to have an interventional radiology procedure for needle-biopsy or radiofrequency ablation purposes in liver or Kidney.
* Only subjects who have provided written informed consent for the study can be included in the study.

Exclusion Criteria:

* Patients have a known allergy to fluorescein
* Patient is Pregnant or breast-feeding
* Patient under judiciary control
* Patient under the tutelage of a guardian
* Patient unable to sign the information consent form (in case of an emergency situation or difficulty in understanding the information)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy (sensitivity specificity) of endomicroscopy as compared to histopathology | up to 2 weeks
  Assessment of the accuracy of Cellvizio confocal mini probe imaging guided by fluoroscopy at the tumor boundary compared with traditional histopathology from physical biopsies

SECONDARY OUTCOMES:
Measure adverse events frequency in the use of mini probes on the tumor | Up to 1 week
  Assessment of the safety of inserting Cellvizio confocal miniprobe in the tumor (nor increase in bleeding or tumor cell dissemination) through the frequency, type and severity of adverse events
Classification of endomicroscopy images from benign and malignant conditions | Up to 6 months
  A first creation of an atlas of endomicroscopic images obtained in interventional radiology with corresponding correlation with traditional pathology images
Percentage of biopsies guided by nCLE (needle-based Confocal Laser Endomicroscopy) which provide a definitive diagnosis as a measure of efficiency of endomicroscopy-targeted biopsies compared to traditional needle biopsies | Up to 5 months
  Yield of nCLE (needle-based confocal laser endomicroscopy)-targeted Fluoroscopy-guided biopsies to assess improvements compared to standard of care from guidance function of the device combination
Number of patients for whom endomicroscopy could have affected the clinical workflow | Up to 5 months
  Evaluation of the potential impact of the endomicroscopic information used in conjunction with the Siemens SOMATOM Definition system in clinical decision-making for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Gangi, Principal Investigator — NHC, Strasbourg, France
Locations (1):
- Nouvel Hôpital Civil, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No